CLINICAL TRIAL: NCT03662204
Title: Blood Sample Collection to Evaluate Biomarkers in Subjects With Untreated Solid Tumors
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-01
Record Dates: First submitted 2018-08-30; First posted 2018-09-07 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Lung Cancer; Colorectal Cancer; Prostate Cancer; Bladder Cancer; Uterine Cancer; Kidney Cancer; Renal Pelvis Cancer; Pancreatic Cancer; Liver Cancer; Stomach Cancer; Ovarian Cancer; Esophageal Cancer
Keywords: blood draw; sample collection
MeSH Terms: conditions — Breast Neoplasms; Lung Neoplasms; Colorectal Neoplasms; Prostatic Neoplasms; Urinary Bladder Neoplasms; Uterine Neoplasms; Kidney Neoplasms; Pancreatic Neoplasms; Liver Neoplasms; Stomach Neoplasms; Ovarian Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Breast: Subjects with clinically confirmed breast cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Lung: Subjects with clinically confirmed lung cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Colorectal: Subjects with clinically confirmed colorectal cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Prostate: Subjects with clinically confirmed prostate cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Bladder: Subjects with clinically confirmed or suspicion of bladder cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Uterine: Subjects with clinically confirmed uterine cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Kidney & Renal Pelvis: Subjects with clinically confirmed or suspicion of kidney or renal pelvis cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Pancreatic: Subjects with clinically confirmed or suspicion of pancreatic cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Liver: Subjects with clinically confirmed liver cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Stomach: Subjects with clinically confirmed stomach cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Ovarian: Subjects with clinically confirmed or suspicion of ovarian cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection
- Esophageal: Subjects with clinically confirmed esophageal cancer and who are treatment naive will provide a blood sample at time of enrollment. No additional blood draws will occur.
  Interventions: Other: Blood Sample Collection

INTERVENTIONS:
Other: Blood Sample Collection — Subjects participating in the study will have blood drawn at enrollment.

SUMMARY:
The primary objective of this study is to obtain de-identified, clinically characterized, whole blood specimens to evaluate biomarkers associated with cancer for diagnostic assay development.

DETAILED DESCRIPTION:
Subjects who have been diagnosed, or who have a suspicion of diagnosis based on imaging, with any solid tumor. Subjects will have a blood sample collected at enrollment and provide medical history prior to initiation of treatment. There will be no further follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female > 18 years of age.
2. Subject has an untreated primary malignancy of breast, lung, colorectal, prostate, bladder, uterine, kidney/renal pelvis, pancreatic, liver, stomach, ovarian or esophageal cancer.

   OR

   Subject has suspicion of a primary malignancy of pancreatic, bladder, kidney/renal pelvis, or ovarian cancer based on imaging.
3. Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Prior or concurrent cancer diagnosis defined as:

   1. Any previous cancer diagnosis within the past 5 years (with the exceptions of basal cell or squamous cell skin cancers); OR
   2. Recurrence of the same primary cancer within any timeframe; OR
   3. Concurrent diagnosis of multiple primary cancers
2. Chemotherapy and/or radiation therapy within 5 years prior to enrollment/sample collection.
3. Any treatment for the primary malignancy or sites of metastases. Subject may not have started neo-adjuvant chemotherapy, neo-adjuvant radiation therapy, immunotherapy or other treatment and/or surgery prior to blood sample collection.
4. Less than 3 days between fine needle aspiration (FNA) of target pathology and blood collection.
5. Less than 7 days between biopsy (other than FNA) of target pathology and blood collection.
6. IV contrast (e.g. CT and MRI) within 1 day [or 24 hours] of blood collection.
7. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 7500 subjects will be enrolled. Subjects will be men and women, 18 years of age and older, who have an untreated breast, lung, colorectal, prostate, bladder, uterine, kidney/renal pelvis, pancreatic, liver, stomach, ovarian or esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 5133 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Biomarker Evaluation | Point in time (one day) blood collection at enrollment
  Biomarkers under evaluation include differential methylation of nucleic acids and altered expression of proteins in blood from subjects with solid tumor cancers.

CONTACTS AND LOCATIONS:
Locations (119):
- United States (119):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Scottsdale Medical Imaging Research, Scottsdale, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Urological Associates of Southern Arizona, PC, Tucson, Arizona
  - Mercy Research-Fort Smith, Fort Smith, Arkansas
  - Genesis Cancer Center, Hot Springs, Arkansas
  - NEA Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - CARTI Cancer Center, Little Rock, Arkansas
  - John Muir Clinical Research, Concord, California
  - Marin Cancer Care, Greenbrae, California
  - Alliance Research Centers, Laguna Hills, California
  - Office of John Homan, MD, Newport Beach, California
  - North County Oncology, Oceanside, California
  - UCI Department of Urology, Orange, California
  - Sharp Memorial Hospital, San Diego, California
  - St. Joseph Heritage Healthcare, Santa Rosa, California
  - Adventist Health - Saint Helena Hospital, St. Helena, California
  - Innovative Clinical Research Institute, Whittier, California
  - RMR VA Medical Center, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Middlesex Hospital, Middletown, Connecticut
  - Easter Ct Hematology and Oncology, Norwich, Connecticut
  - Stamford Hospital, Stamford, Connecticut
  - Southeast Florida Hematology-Oncology Group, PA, Fort Lauderdale, Florida
  - CSNF - Central Business Office, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Piedmont Cancer Institute, PC, Atlanta, Georgia
  - Candler Hospital, Savannah, Georgia
  - Lewis Hall Singletary Oncology Center, Thomasville, Georgia
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - PMG Research of DuPage Medical Group, Downers Grove, Illinois
  - Presence Cancer Care / JOHA, Joliet, Illinois
  - Illinois CancerCare, P.C., Peoria, Illinois
  - Orchard Healthcare Reasearch Inc, Skokie, Illinois
  - SIU School of Medicine, Springfield, Illinois
  - Investigative Clinical Research of Indiana, LLC, Indianapolis, Indiana
  - PMG Research of McFarland Clinic, Ames, Iowa
  - Des Moines Oncology Research Associate, Des Moines, Iowa
  - Oncology Fort Thomas St. Elizabeth's Edgewood Cancer Care Research, Edgewood, Kentucky
  - Baptist Health-Lexington, Lexington, Kentucky
  - Norton Cancer Institute-Pavilion, Louisville, Kentucky
  - Baptist Health, Louisville, Kentucky
  - Baptist Health- Paducah, Paducah, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Holy Cross Hospital Resource Center Department of Cancer Research, Silver Spring, Maryland
  - Beverly Hospital, Oncology, Beverly, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Cancer and Hematology Centers of Western Michigan, PC, Grand Rapids, Michigan
  - Cancer Research Consortium of West Michigan (CRCWM), Grand Rapids, Michigan
  - Ascension Providence Hospitals, Southfield, Michigan
  - Metro-Minnesota Community Oncology Research Consortium (MMCORC), Saint Louis Park, Minnesota
  - Park Nicollet Institute - Oncology Research, Saint Louis Park, Minnesota
  - St. Dominic's Gynecologic Oncology, Jackson, Mississippi
  - North Mississippi Medical Center Hematology and Oncology, Tupelo, Mississippi
  - Mercy Cancer Center, Joplin, Missouri
  - Mercy Cancer and Hematology Clinic, Springfield, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Nebraska Hematology-Oncology -- Lincoln, Lincoln, Nebraska
  - Somnos Laboratories, Inc., Lincoln, Nebraska
  - Cancer Care Specialists, Reno, Nevada
  - The Minniti Center for Hematology and Oncology, Mickleton, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Albany Medical College, Albany, New York
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York, East Syracuse, New York
  - Premier Medical Group of the Hudson Valley PC, Poughkeepsie, New York
  - Premier Medical Group of the Hudson Valley, PC Research Department - Gastroenterology Division, Poughkeepsie, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook Cancer Center, Stony Brook, New York
  - Associated Medical Professionals, Syracuse, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - PMG Research of Piedmont, Statesville, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Zimmer Cancer Center, Wilmington, North Carolina
  - Hematology & Oncology Associates, Inc., Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Inc., Massillon, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Genie Jackson Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Mercy Oncology Research, Oklahoma City, Oklahoma
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Charleston Cancer Center, Charleston, South Carolina
  - McLeod Center for Cancer Treatment and Research, Florence, South Carolina
  - Saint Francis Cancer Center Research Department, Greenville, South Carolina
  - Lowcountry Urology/PMG Research of Charleston, LLC, North Charleston, South Carolina
  - Spartanburg Medical Center: Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - RH Clinical Research, Rapid City, South Dakota
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - The Jackson Clinic, Jackson, Tennessee
  - Christus Spohn Cancer Center, Corpus Christi, Texas
  - University of Texas Health Science Center, Houston, Texas
  - Sun Research Institute, San Antonio, Texas
  - San Antonio Military Medical Center, San Antonio, Texas
  - Cancer Treatment Center, Texarkana, Texas
  - Renovatio Clinical, The Woodlands, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Urology of Virginia, PLLC, Virginia Beach, Virginia
  - Seattle Urology Research Center, Burien, Washington
  - MultiCare Regional Cancer Center, Tacoma, Washington
  - CAMC Clinical Trials Center, Charleston, West Virginia
  - Mon Health Medical Center, Morgantown, West Virginia
  - West Virginia University Cancer Institute, Morgantown, West Virginia
  - HSHS St. Vincent Hospital, Green Bay, Wisconsin
  - Michael Berry Building-Oncology, Janesville, Wisconsin
  - UW Carbone Cancer Center, Madison, Wisconsin
  - ProHealth Care Research Institute, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study will be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol and informed consent form (when applicable) will also be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available from 2 years and ending 4 years after publication. Data will be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.